CLINICAL TRIAL: NCT06408506
Title: In-patient Comparison of Immediately Loaded and Non-loaded Submerged and Transgingival Healed Implants Within 4 Months A Controlled Clinical Pilot Study
Brief Title: In-patient Comparison of Immediately Loaded and Non-loaded Submerged and Transgingival Healed Implants Within 4 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29-172 ex 16/17
Record Dates: First submitted 2024-04-29; First posted 2024-05-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Jaw, Edentulous
Keywords: Immediate loading; Prei-implant bone regeneration; Implant Survival
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Masking Description: The positioning and loading protocols of the implants under investigation are blinded to the investigator during the analysis of peri-implant bone heights, which are measured using periodontal probes, as well as during the analysis of intraoperative scans and impressions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6 Implants in edentulous mandible (Other): Placement of 6 Implants in the lower jaw, Two of which are remained to heal submucosal, two transmucosal, and two by immediate loading with removable gold bar retained dentures
  Interventions: Procedure: Re-Entry Surgery; Procedure: Probing peri-implant bone; Procedure: Scanning peri-implant bone; Procedure: Conventional Impressions; Procedure: Implant Surgery; Procedure: Healing procedure

INTERVENTIONS:
Procedure: Re-Entry Surgery — Re-entry surgery 4 months after the insertion of the implants to reveal implants after osseointegration
Procedure: Probing peri-implant bone — Probing peri-implant bone with Dental Probe during surgery
Procedure: Scanning peri-implant bone — Scanning peri-implant bone during surgery
Procedure: Conventional Impressions — Conventional Impressions during surgery
Procedure: Implant Surgery — Placement of 6 implants in the edentulous mandible
Procedure: Healing procedure — All 6 Implants in all patients are let to heal for 4 Months under the same conditions:
  The most distal implants are left submerged. The most mesial implants are left transgingival and the Implants in the middle are immediately loaded using gold bar retained dentures

SUMMARY:
The study involves 20 patients who require implant treatment for the edentulous lower jaw, following specific inclusion and exclusion criteria. Patients are drawn from the regular pool of those seeking implant therapy, with no additional recruitment efforts.

This study compares the effects of loaded and non-loaded dental implants. Preoperative assessments include medical histories, clinical, and radiographic examinations of the jaw. Participants are thoroughly informed about the study procedures and consent to participate through signed agreements. They undergo preoperative diagnostics, including panoramic X-rays to evaluate mandibular bone height, and complete the OHIP-G 14 questionnaire to establish a baseline for their oral health-related quality of life.

The implant placement involves standard outpatient surgical procedures under local anesthesia. The implants used are CE-certified and are placed in predetermined positions in the edentulous region. During the surgery intraoral scans and conventional impressions are performed. Post-operative care includes oral rinses, and radiographic assessments, with follow-up visits scheduled for suture removal and further assessments using the visual analog scale for pain and swelling.

The healing phase spans four months, during which patients' comfort and oral health are monitored through clinical examinations and additional questionnaires. Follow-up after 4 months includes re-entry surgery and further radiographic evaluations and intraoral scans to assess the bone's response around the implants. Throughout the study, adverse events and patient satisfaction are continuously documented.

In the later stages, regular follow-up visits for up to 24 months post-surgery to monitor implant stability and health through clinical and radiographic check-ups are performed.

This study aims to document implant survival rates, peri-implant bone regeneration, assess biological and technical complications, and evaluate patient satisfaction and quality of life throughout the implant process, providing valuable data for future dental implant protocols.

DETAILED DESCRIPTION:
The clinical study conducted at the Dental School of the Medical University of Graz is designed to evaluate the effects and outcomes of loaded versus non-loaded dental implants in patients requiring treatment for an edentulous lower jaw. This study includes 20 patients who meet specific inclusion and exclusion criteria and are recruited from the regular pool of patients at the facility, without any special recruitment efforts.

Study Overview The primary objective of this study is to compare the integration and performance of loaded and non-loaded dental implants. Before the study procedures begin, each participant undergoes a thorough preoperative evaluation, which includes a complete medical history review and a detailed clinical and radiographic examination of the recipient site in the jaw. These initial assessments are crucial for ensuring patient safety and suitability for the study.

Informed Consent and Patient Information All participants receive detailed patient information leaflets that explain the study's purpose, procedures, potential risks, and benefits. This is followed by obtaining informed consent through a separate agreement form, ensuring that all participants are fully aware and agreeable to the study's terms.

Preoperative Procedures The preoperative phase includes radiological diagnostics, such as panoramic x-rays to evaluate the mandibular bone and measure residual bone height. Additionally, participants complete the OHIP-G 14 questionnaire to gauge their oral health-related quality of life at baseline. Intraoral photographs are also taken to document each patient's initial condition.

Surgical Procedure and Implant Placement The surgical procedures are performed under local anesthesia in a septic environment typical of outpatient settings. Each patient rinses with a 0.2% chlorhexidine digluconate solution preoperatively. A full-thickness flap is prepared, and the bone is assessed for quality and quantity before implant placement. The implants, all CE-certified and of the same design, are placed in six predetermined positions in the interforaminal region of the lower jaw.

Postoperative Care and Assessments After implant placement, excessive bleeding is controlled, and the surgical site's condition is documented with intraoperative photographs and radiographs. Probing to assess the peri-implant bone height is applied, as well as intraoral scanning and conventional impressions are performed. A panoramic x-ray and individual x-rays of the implants are taken immediately post-surgery. The implants placed are either immediately loaded with a rotating gold bars or left to heal submerged or transgingival based on their predetermined positions. Postoperative care includes prescribing antibiotics and anti-inflammatory medications as necessary, and the administration of these drugs is meticulously documented.

Follow-up Visits and Ongoing Evaluations The follow-up phase includes several visits where the integration of the prosthetic components to the loaded implants is assessed and sutures are removed. The patients' perceptions and acceptance of the implant and prosthetic fit are evaluated using a visual analog scale for pain and swelling. The quality of life is continuously monitored through repeated administration of the OHIP-G 14 questionnaire.

Healing Period A four-month healing period follows, during which the implants are monitored through regular clinical checks. These include sensitivity tests, patient comfort tests, and evaluations of general patient satisfaction.

Secondary Surgery and Long-Term Follow-up A secondary surgery for exposing the remaining implants, assessment of peri-implant bone remodeling using periodontal probes and intraoral scans as well as conventional impressions and further radiographic and clinical assessments are scheduled. The study concludes with long-term follow-up visits, which include professional tooth cleaning and routine check-ups to monitor the implants' stability and the peri-implant conditions.

Data Collection and Analysis Throughout the study, data is collected on implant survival rates, incidence of biological and technical complications, and patient satisfaction. Standardized periapical and panoramic radiographs are taken at various stages to serve as routine clinical assessments, and a detailed scan analysis is performed to document bone quantity changes around the implants.

Conclusion This comprehensive study aims to provide valuable insights into the comparative effectiveness of loaded and non-loaded implants, contributing to the optimization of treatment protocols for dental implant therapy. Through meticulous documentation and rigorous follow-up, the study seeks to enhance understanding of the factors that influence implant success and patient satisfaction, ultimately improving outcomes in dental implantology.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the participant after being informed Capability of giving an informed consent
* good health as defined by the subjects medical history (no contraindications as described in the exclusion criteria below)
* age 20 to 80 years
* Patients who require 6 implants in the positions 32, 33, 34, 42, 43, 44
* edentulous mandible with enough interforaminal bone volume for placement of 6 implants
* Residual vertical bone height of at least 8mm in the interforaminal region
* Patients who wish implant-supported restoration with six implants

Exclusion Criteria:

* Homelessness
* Smoking
* Medication with a contraindication for implant therapy
* Skeletal immaturity
* Any active malignancy or ongoing treatment for malignancy
* An active infection at the operative site
* Persistent compartment syndrome or neurovascular residua of compartment syndrome
* Pathological fractures such as those observed in (but not limited to) Paget's disease or in metastatic bone
* Contraindications to the class of devices under study, e.g. known hypersensitivity or allergy to class of devices
* Pregnancy
* Intention to become pregnant during the course of the study
* Breast feeding
* Lack of safe contraception

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Survival | 24 months
  Implant survival

SECONDARY OUTCOMES:
Peri-implant bone height | 0 and 4 months
  Bone heights assessed using probing, and by digitally measuring intraoperative impressions.
Oral Health Impact Profile-14 in German | 0 to 24 months
  The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. The domain scores can range from 0 to 8. Higher OHIP-14 scores indicate worse and lower scores indicate better Oral Health Related Quality of Life
Bleeding on Probing | 0 to 24 months
  Bleeding on probing is a simple and accurate indicator of the health of the peri-implant tissues. The presence or degree of peri-implant mucositis can be associated by the degree of bleeding and the possibility of progression into peri-implantitis.The ideal soft tissue condition around an implant is an absence of BOP
Plaque Index | 0 to 24 months
  Clinical plaque index is used to evaluate the level and rate of plaque formation on prosthetic surface, and to monitor the patients' dental hygiene. A "good" plaque Index is considered between 0.3- 0.6; as "fair" when it is 0.7 - 1.8; or "poor" when the score is between 1.9 to 3.0.
Probing Around Implants | 0 to 24 months
  Probing periimplant pocket depths for peri-implant monitoring. Long-term clinical investigations have shown that desirable probing depths around dental implants are 2.5mm to 4mm, but deeper assessments can also be associated with healthy peri-implant mucosa.
Visual Analogue Scale for Pain assessment | 0 to 24 months
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). The patient is asked to rate their current level of pain by placing a mark on the line.

CONTACTS AND LOCATIONS:
Overall Officials: Alwin Sokolowski, DDS,MDS,PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Dental Department Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorenzoni M, Pertl C, Zhang K, Wegscheider WA. In-patient comparison of immediately loaded and non-loaded implants within 6 months. Clin Oral Implants Res. 2003 Jun;14(3):273-9. doi: 10.1034/j.1600-0501.2003.140304.x. PMID 12755777
- [Background] Ericsson I, Randow K, Nilner K, Peterson A. Early functional loading of Branemark dental implants: 5-year clinical follow-up study. Clin Implant Dent Relat Res. 2000;2(2):70-7. doi: 10.1111/j.1708-8208.2000.tb00108.x. PMID 11359266
- [Background] Siddiqui AA, Ismail JY, Kukunas S. Immediate loading of dental implants in the edentulous mandible: a preliminary case report from an international prospective multicenter study. Compend Contin Educ Dent. 2001 Oct;22(10):867-70, 873-4, 876 passim; quiz 884. PMID 11915636
- [Background] Schulte W, Lukas D. Periotest to monitor osseointegration and to check the occlusion in oral implantology. J Oral Implantol. 1993;19(1):23-32. PMID 8246291
- [Derived] Sokolowski A, Lorenzoni M, Steyer E, Marschner F, Pichler A, Sokolowski A. In-patient comparison of marginal bone loss after 4 months in immediately loaded, submucosal, and transmucosal dental implants using 3D scanning: a prospective clinical trial. Clin Oral Investig. 2025 Mar 17;29(4):186. doi: 10.1007/s00784-025-06255-y. PMID 40095138

DOCUMENTS (1):
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT06408506/Prot_000.pdf